CLINICAL TRIAL: NCT07002710
Title: Impact of Persistent Inflammation-Immunosuppression-Catabolism Syndrome (PICS) on the Respiratory Physiology in Patients With Prolonged Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407047RINE
Record Dates: First submitted 2024-12-26; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: PICS
Keywords: PICS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Past research on PICS has mainly focused on the predictability and prognosis of PICS occurrence in ICU patients. Still, there is currently insufficient research on the role of PICS in the care setting of patients who have stabilized and are transferred to respiratory care units such as Respiratory Care Centers (RCCs) for weaning attempts. To understand the impact of PICS on the respiratory physiology of patients undergoing weaning from prolonged mechanical ventilation, investigators propose a one-year research plan

DETAILED DESCRIPTION:
Past research on PICS has mainly focused on the predictability and prognosis of PICS occurrence in ICU patients. Still, there is currently insufficient research on the role of PICS in the care setting of patients who have stabilized and are transferred to respiratory care units such as Respiratory Care Centers (RCCs) for weaning attempts. To understand the impact of PICS on the respiratory physiology of patients undergoing weaning from prolonged mechanical ventilation, investigators propose a one-year research plan with the hypothesis that PICS endotype patients in the RCC setting are more likely to develop alveolar collapse during weaning trials, leading to decreased oxygenation function, increased respiratory burden, and potentially more lung injury from repeated alveolar collapse and reopening. Investigators plan to enroll 60 PMV patients admitted to the RCC, perform laboratory analyses to categorize patients as PICS endotype or other types, and then collect clinical data, respiratory physiology data, and biomarkers during weaning trials, such as changes in oxygenation, respiratory work and energy expenditure, infection occurrence, diaphragm ultrasound, esophageal pressure measurements, electrical impedance tomography, and inflammatory biomarkers. The expected research outcomes include the prevalence of PICS in stable PMV patients in the RCC setting and the differences in respiratory physiology and weaning outcomes between PICS and non-PICS patients, which could inform differentiated or personalized weaning strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients are still receiving ventilator support when transferred to the ward where the study is conducted.
* Use the respirator continuously for at least 10 days.
* Vital signs are stable: blood pressure systolic blood pressure is not lower than 70 mmHg; heartbeat is not lower than 50/min and not higher than 160/min; respiratory rate is not higher than 50/min.
* When using respirator support, the oxygen concentration should not exceed 60%.

Exclusion Criteria:

．At least one of the following conditions occurs: 1. Pregnancy. 2. The patient refuses to undergo weaning from the respirator training. 3. The patient has no ability to drive spontaneous breathing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential candidates for screening are adult patients transferred from RCC who are still on ventilators and will undergo screening assessment by researchers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Persistent Inflammation-Immunosuppression-Catabolism Syndrome (PICS) on the Respiratory Physiology in Patients with Prolonged Mechanical Ventilation | January 1st,2025 to December 31st,2026
  To understand whether weaning training strategies for PICS and non-PICS patients may have different considerations when patients undergo spontaneous breathing testing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan